CLINICAL TRIAL: NCT00382824
Title: Effects of Coenzyme Q10 in Progressive Supranuclear Palsy (PSP): A Multicenter, Randomized, Placebo-controlled, Double Blind Study
Brief Title: Effects of Coenzyme Q10 in Progressive Supranuclear Palsy (PSP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LaheyC
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-06

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive Supranuclear Palsy; CoQ10; Coenzyme Q10
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — coenzyme Q10

STUDY DESIGN:
Intervention Model Description: Multicenter, Double-blind, Randomized, Placebo-Controlled Clinical Trial to examine tolerability, safety, and efficacy of CoenzymeQ10
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CoQ10 (Active Comparator): Half of the enrolled patients will be randomized into the the CoQ10 arm and will receive a dosage of 2400mg/day of Coenzyme Q10
  Interventions: Dietary Supplement: Coenzyme Q10
- Placebo (Placebo Comparator): Half of the enrolled patients will be randomized into the the Placebo arm and will receive a matching dose of placebo that resembles the 2400mg/day dose of the CoQ10 arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — active drug
  Other Names: CoQ10
  Arms: CoQ10
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The clinical syndrome of PSP responds poorly to all available forms of therapy used in Parkinson's Disease (PD). Currently, no effective treatment exists. Coenzyme Q10 in high doses has been shown to be a beneficial therapy in PD and might possibly be a beneficial therapy for PSP. This study will compare the efficacy, safety and tolerability of Coenzyme Q10 versus placebo in patients with atypical parkinsonian syndrome, progressive supranuclear palsy (PSP).

DETAILED DESCRIPTION:
The study is designed as a multicenter randomized, placebo-controlled, double blind trial. Up to 60 patients with PSP will be enrolled at several centers in the United States

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the diagnostic criteria of PSP/diagnosed within the past 5 years
* Either vertical supranuclear palsy or both slowing of vertical saccades
* Prominent postural instability with falls in the first year of disease onset
* No evidence of other diseases that could explain the foregoing features

Exclusion Criteria:

* Current or previous therapeutic use of CoQ10
* Parkinsonism due to drugs
* History of pallidotomy, thalamotomy, active deep brain stimulator or fetal tissue transplant
* History of active epilepsy, stroke, structural brain disease
* Use of methylphenidate hydrochloride, cinnarizine, reserpine, amphetamines, or monoamine oxidase-A inhibitors within 3 months before the baseline visit.
* Active cancer or cancer undergoing treatment
* Participation in other drug studies or the use of other investigational drugs within 30 days before screening.
* Known hypersensitivity to Coenzyme Q10.
* Pregnant, planning a pregnancy or nursing woman

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-09; Primary Completion 2013-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Apetauerova, MD, Principal Investigator — Lahey Clinic
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Apetauerova D, Scala SA, Hamill RW, Simon DK, Pathak S, Ruthazer R, Standaert DG, Yacoubian TA. CoQ10 in progressive supranuclear palsy: A randomized, placebo-controlled, double-blind trial. Neurol Neuroimmunol Neuroinflamm. 2016 Aug 2;3(5):e266. doi: 10.1212/NXI.0000000000000266. eCollection 2016 Oct. PMID 27583276
- See also: CurePSP homepage — http://www.psp.org
- See also: Lahey Clinic homepage — http://www.lahey.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Coenzyme Q10 (2400mg/Day): Patients randomized into this arm received 2400mg of coenzyme Q10 per day (300mg wafers eight times per day). Each wafer also contained 200IU of vitamin E for a total of 1200IU of vitamin E/day. Patients in this group were to take this dose for 12 months.
- Placebo: Patients randomized into this arm received placebo wafers. These wafers looked identical to the Coenzyme Q10 wafers. Patients took 8 placebo wafers per day. Each wafer also contained 200IU of vitamin E. Patients received 1200IU of viatmin E/day
Period: Overall Study
Arm/Group | Coenzyme Q10 (2400mg/Day) | Placebo
Started | 32 | 29
Completed | 20 | 16
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Coenzyme Q10 (2400mg/Day): Patients randomized into this arm received 2400mg of coenzyme Q10 per day (300mg wafers eight times per day). Each wafer also contained 300IU of vitamin E. Patients in this group were to take this dose for 12 months.
- Placebo: Patients randomized into this arm received placebo wafers. These wafers looked identical to the Coenzyme Q10 wafers. Patients took 8 placebo wafers per day.
- Total: Total of all reporting groups
Arm/Group | Coenzyme Q10 (2400mg/Day) | Placebo | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Customized [Mean (Full Range); unit: years] — cannot edit Baseline Measure Title
  years
    Age | 66.3 [32 to 89] | 66.9 [53 to 85] | 66.6 [32 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 24
  Male | 24 | 13 | 37

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Coenzyme Q10 (Unified Parkinson's Disease Rating Scale [UPDRS] AND Progressive Supranuclear Palsy Rating Scale [PSPRS])
Description: Unified Parkinson's Disease Rating Scale [UPDRS]: Higher scores indicate a higher degree of impairment The total score is calculated by summing the subscores. Total scores range from 0 (normal) to 166 (severely impaired) Part I [Mentation, Behavior, & Mood] Scale: 0-16 Part II [Activities of Daily Living, Both "ON" & "OFF"] Scale:0-52 Part III [Motor Examination] Scale: 0-56 Part IV [Complications of Therapy] Scale: 0-34 Part V [Modified Hoehn & Yahr Staging] Scale: 0-8 Part VI [Schwab & England Activities of Daily Living Scale] Scale: 0 - 100%
  Progressive Supranuclear Palsy Rating Scale [PSPRS] - Total Scale ranges from 0 (normal) to 128 (severely impaired) Section 1 [History] Scale: 0-31 Section 2 [Mentation] Scale: 0-20 Section 3 [Bulbar] Scale: 0-10 Section 4 [Ocular Motor] Scale: 0-20 Section 5 [Limb Motor] Scale: 0-22 Section 6 [Gait and midline] Scale: 0-25
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coenzyme Q10 (2400mg/Day) | Placebo
Number analyzed (Participants) | 20 | 16
units on a scale
  Change in UPDRS scores | 5.9 (10.0) | 11.8 (8.6)
  Change in PSPRS scores | 11.5 (11.1) | 12.8 (9.1)

2. Secondary Outcome: Efficacy of Coenzyme Q10 (Mini-Mental State Examination [MMSE] and Activities of Daily Living [ADL] Scales)
Description: Efficacy of Coenzyme Q10 measured by change in intellectual function (the Mini-Mental State Examination [MMSE]) and Activities of Daily Living (ADL) scores.
  MMSE: 30 point scale with 5 subsections (Total Score Range: minimum score = 0, maximum = 30): Orientation (max=10 pts, min=0 pts), Registration (max=3 pts, min=0 pts), Attention & Calculation (max=5pts, min=0 pts), Recall (max=3 pts, min= 0 pts), Language & Praxis (max=9 pts, min=0 pts). Lower scores indicate greater impairment. Scores <24 are considered abnormal.
  Activities of Daily Living scores:
  The UPDRS part II is used to assess subject's degree in which they can perform their Activities of Daily Living. Part II of the UPDRS rates subjects on a 0-4 scale, with 0 being "Normal" and 4 being "Severe Impairment", for each respective item. For each item, the reported score is divided by the maximum total score for that item and multiplied by 100 to give a 0-100 scale range. Higher scores indicate greater impairment.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coenzyme Q10 (2400mg/Day) | Placebo
Number analyzed (Participants) | 20 | 16
units on a scale
  Change in ADL scores | -13.5 (20.6) | -18.4 (15.9)
  Change in MMSE scores | -1.3 (3.4) | -1.3 (1.8)

3. Secondary Outcome: Quality of Life Questionnaires: Parkinson's Disease Questionnaire - 39 [PDQ-39], Short Form-36 [SF-36]
Description: Parkinson's Disease Questionnaire - 39 (PDQ-39): 39 Items. 8 subscales: mobility, activities of daily living, emotional well-being, stigma, social support , cognitions, communication, bodily discomfort. Subjects indicate never (0 pts), occasionally (1 pts), sometimes (2pts), often (3pts), or always/cannot do at all (4pts) for each item in each section. The sum of scores of each item in the dimension divided by the maximum possible score of all the items in the dimension, multiplied by 100. Range of scores for each dimension: 0-100. The sum of dimension total scores are divided by 8 to calculate the Parkinson's Disease Severity Index. Range of total score for the Parkinsons' Disease Severity Index: 0-100. Lower scores indicate better quality of life.
  Short Form-36 (SF-36): 36 items 8 subscales: (2) General Health Sections, Limitations of Activities, Physical Health Problems, Emotional Health Problems, Pain, (2) Social Activities sections, and Energy and Emotions. Each qu
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coenzyme Q10 (2400mg/Day) | Placebo
Number analyzed (Participants) | 20 | 16
units on a scale
  Change in Parkinson's Disease Questionnaire scores | 3.4 (13.9) | 7.5 (12.6)
  Change in Short Form-36 Scores | -2.1 (19.1) | -7.2 (15.4)

4. Secondary Outcome: Safety Profile of Coenzyme Q10
Description: The safety Profile of Coenzyme Q10 as determined by the analysis of the frequency and severity of the adverse event data, changes in the vital signs, electrocardiograms and clinical laboratory values, recorded over the course of the trial.
Time Frame: 12 months
Measure: Number; unit: Adverse Events
Arm/Group | Coenzyme Q10 (2400mg/Day) | Placebo
Number analyzed (Participants) | 32 | 29
Adverse Events
  Adverse Events | 27 | 38
  Serious Adverse Events | 5 | 8

5. Secondary Outcome: Tolerability of Coenzyme Q10
Description: 1. The tolerability of Coenzyme Q10 as determined by the number of subjects who complete the study on their original treatment assignment, and
  2. The tolerability of Coenzyme Q10 as determined by the number of subjects completing the study.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Coenzyme Q10 (2400mg/Day) | Placebo
Number analyzed (Participants) | 32 | 29
Participants | 20 | 16

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Coenzyme Q10 (2400mg/Day) | Placebo
Serious Adverse Events (participants affected / at risk) | 5/32 | 8/29
Other Adverse Events (participants affected / at risk) | 11/32 | 8/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coenzyme Q10 (2400mg/Day) (N=32) | Placebo (N=29)
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Aspiration pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Benign postatic hyperplasia with obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Stent placement (Surgical and medical procedures) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
C. difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Bleeding ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ureteral calculus (Renal and urinary disorders) | 0 (0) | 1 (1)
Laceration to head (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coenzyme Q10 (2400mg/Day) (N=32) | Placebo (N=29)
Urinary tract infection (Renal and urinary disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Cataract (Eye disorders) | 2 (2) | 1 (1)
Nausea (General disorders) | 2 (2) | 1 (1)
Diarrhea (General disorders) | 2 (2) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No